CLINICAL TRIAL: NCT01053481
Title: Using Ca-41 Methodology to Assess the Impact of Different Vitamin D Supplementation Levels on Postmenopausal Bone Health
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof. Dr. med, Swiss Federal Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2009-04-07-Ca41
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vitamin D (Experimental): Vitamin D supplement
  Interventions: Dietary Supplement: vitamin D; Behavioral: exercise program (rebounding on a trampoline)

INTERVENTIONS:
Dietary Supplement: vitamin D — Vitamin D supplement
Behavioral: exercise program (rebounding on a trampoline) — 40 days at 30 min/d

SUMMARY:
The purpose of this study is to determine whether increasing levels of serum 25(OH)Vitamin D as achieved by oral supplementation higher than the current recommendations are associated with a less negative bone calcium balance in post-menopausal Swiss women.

DETAILED DESCRIPTION:
In a substudy - not related to the vitamin D intervention - spot and 24 h urine samples are compared with regard to the assessment of iodine status in Swiss post-menopausal women.

In an short subsequent study using five of the subjects who participated in the original trial, the effect of a 40 d-exercise program (rebounding on a trampoline) on Ca-41 excretion will be observed.

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy women, at least 5 years post-menopausal
* BMI 18-30
* no HRT
* no regular intake of Ca or vit D supplements
* wiling and able to give written informed consent and to understand, participate and comply with study requirements
* non-smokers
* no long travels (>3 wk) planned within study period

Exclusion Criteria:

* diseases that predispose to osteoporosis
* history of fragility fractures
* currently on a weight reduction program
* excessive physical activity
* diseases influencing calcium metabolism (thyroid, parathyroid, adrenal disorders etc.)
* regular intake of medication affecting calcium metabolism
* osteoporosis (T-score below -2.5)
* history of psychological illness likely to interfere with the subject's ability to understand the requirements of the study
* participation in concurrent studies

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
urinary Ca-41/Ca-40 ratio | March 2010 to January 2011

SECONDARY OUTCOMES:
biomarkers of bone metabolism | March 2010 to January 2011
urinary iodine | August 2009 to December 2010
  Comparison of spot and 24 h urine samples for the assessment of iodine status (substudy, not related to vitamin D intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zimmermann, Prof. Dr. med., Principal Investigator — ETH Zurich
Locations (1):
- Human Nutrition Laboratory, Institute of Food, Nutrition and Health, ETH Zurich, Zurich, Switzerland

REFERENCES:
- [Background] Denk E, Hillegonds D, Hurrell RF, Vogel J, Fattinger K, Hauselmann HJ, Kraenzlin M, Walczyk T. Evaluation of 41calcium as a new approach to assess changes in bone metabolism: effect of a bisphosphonate intervention in postmenopausal women with low bone mass. J Bone Miner Res. 2007 Oct;22(10):1518-25. doi: 10.1359/jbmr.070617. PMID 17576167
- [Background] Denk E, Hillegonds D, Vogel J, Synal A, Geppert C, Wendt K, Fattinger K, Hennessy C, Berglund M, Hurrell RF, Walczyk T. Labeling the human skeleton with 41Ca to assess changes in bone calcium metabolism. Anal Bioanal Chem. 2006 Nov;386(6):1587-602. doi: 10.1007/s00216-006-0795-5. Epub 2006 Oct 11. PMID 17033771
- [Derived] Schild A, Herter-Aeberli I, Fattinger K, Anderegg S, Schulze-Konig T, Vockenhuber C, Synal HA, Bischoff-Ferrari H, Weber P, von Eckardstein A, Zimmermann MB. Oral Vitamin D Supplements Increase Serum 25-Hydroxyvitamin D in Postmenopausal Women and Reduce Bone Calcium Flux Measured by 41Ca Skeletal Labeling. J Nutr. 2015 Oct;145(10):2333-40. doi: 10.3945/jn.115.215004. Epub 2015 Sep 2. PMID 26338885